CLINICAL TRIAL: NCT04131504
Title: A Multi-Center, Prospective Study to Discover a Companion Diagnostic for Biologics Targeting TNF
Brief Title: Precision Crohn's Disease Management Utilizing Predictive Protein Panels (ENvISION)
Acronym: ENvISION
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0730
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Crohn's Disease; IBD
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood specimens will be collected for biomarker discovery and validation
  * Stool specimens will be collected for microbial analysis and additional IBD-related stool biomarkers
  * OPTIONAL: Four additional research-only intestinal pinch biopsies at the time of a clinically indicated or research-only colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Phase I - Cross-sectional Study (CD and Suspected IBD): 150 children and young adults who have been previously diagnosed with CD (anti-TNF naïve) or suspected of having IBD (based on clinical symptoms and laboratory testing) who are scheduled for a clinically-indicated colonoscopy are eligible to be enrolled in this cohort.
- Phase I - Cross-sectional Study (healthy volunteers): 20 healthy controls will be enrolled at Cincinnati Children's Hospital only. Once demographics, past medical/surgical history and biospecimens (blood/stool) are collected, controls will complete participation.
- Phase II - Longitudinal Study of Participants with CD: 70 children and young adults who have been diagnosed with CD (anti-TNF naïve) and are scheduled to receive infliximab (or adalimumab) are eligible to be enrolled in this cohort.
  Interventions: Drug: Infliximab; Drug: Adalimumab

INTERVENTIONS:
Drug: Infliximab — No standard dosing regimen will be used and the dose will be determined by the treating physician
  Other Names: Remicade
  Groups: Phase II - Longitudinal Study of Participants with CD
Drug: Adalimumab — No standard dosing regimen will be used and the dose will be determined by the treating physician
  Other Names: Humira
  Groups: Phase II - Longitudinal Study of Participants with CD

SUMMARY:
Crohn's disease and ulcerative colitis affect about 1.6 to 3 million people in the United States with many of those being young children and adolescents. Physicians need better ways to inform decisions on therapy selection and recognize ongoing intestinal injury while on treatment.

The main reason for this research study is to see if a blood test or stool test, which measures specific proteins, taken just before starting a new treatment for Crohn's disease can predict a patient's ability to achieve complete intestinal healing. The investigators also want to see if the intensity of gut inflammation can be detected by measuring a separate set of proteins in the blood.

DETAILED DESCRIPTION:
Despite the heterogeneity of CD phenotypes and a potentially aggressive course of inadequately treated CD, treatment selection for newly diagnosed patients is currently based on clinical factors which do not define CD sub-types. Now, with additional biologic therapies for CD, there is a critical need for individual biochemical analysis both pre-treatment, and following induction to assess the probability of durable remission. These data will inform decisions on continued dosing of the current biologic, or whether addition of combination therapy or switching to a therapy with an alternative mechanism of action will be more beneficial.

The Food & Drug Administration (FDA) defines a companion diagnostic as a device that can identify patients most likely to benefit from a therapy or a device to monitor response with the purpose to adjust the treatment to achieve improved effectiveness.Our global aim is to develop a companion diagnostic (peripheral blood panel) that accurately predicts the probability of deep remission (clinical remission with MH) to anti-TNF and a protein (blood) biomarker panel that reproducibly distinguishes endoscopic MH from active (ulcerated) intestinal inflammation in patients with CD.

The long-term strategy is to utilize the "low-risk" anti-TNF specific module (protein panel) to personalize CD therapy. With the addition of new biologics for CD, patients with a low-risk inflammatory profile would not only be expected to achieve MH but also predicted to respond to treatment escalation strategies while avoiding or stopping the drug (if drug exposure is optimized) sooner in patients in which the protein profile predicts a low probability of deep remission with anti-TNF. As additional therapies are approved for pediatric CD, the priority would be to avoid anti-TNF in patients with a "high-risk" protein profile and specifically select therapies that target the patient's individual inflammatory signature. Additionally, the investigators expect the protein profile of patients failing to achieve deep remission to provide further insight into molecular mechanisms contributing to the continued inflammation and thereby directing the next therapeutic option.

ELIGIBILITY:
Phase I - Cross-sectional Study (CD and Suspected IBD)

Inclusion Criteria:

1. Age criteria: > 1 year to < 22 years of age
2. Diagnosis of Crohn's disease, anti-TNF naïve, and colonoscopy scheduled OR
3. Clinical suspicion for IBD (treatment naïve) and colonoscopy scheduled
4. Permission of parent/guardian and assent or consent of research participant

Exclusion Criteria:

1. Any prior treatment with an anti-TNF, such as infliximab, adalimumab, certolizumab or golimumab
2. Known diagnosis of ulcerative colitis (UC) or inflammatory bowel disease-unspecified (IBD-U)
3. Active or prior evidence of internal (abdominal/pelvic) penetrating fistula(e)
4. Active intra-abdominal abscess or perianal abscess
5. Active Clostridium difficile infection or other known enteric infection in last 2 weeks
6. Current ileostomy or colostomy, extensive small bowel resection, ileoanal pouch or short bowel syndrome
7. History of autoimmune disease (including autoimmune hepatitis, primary sclerosing cholangitis, thyroiditis, psoriasis or juvenile idiopathic arthritis)
8. Any condition that in the opinion of the PI will prevent the research participant from taking part in this study

Phase I - Cross-sectional Study (healthy volunteers)

Inclusion Criteria:

1. Age criteria: > 1 year to < 22 years of age
2. Any CCHMC patient
3. Permission of parent/guardian and assent or consent of research participant

Exclusion Criteria:

1. Known diagnosis of one or more of the following: irritable bowel syndrome, gastroesophageal reflux, constipation, BMI>95% for age, small intestinal bacterial overgrowth (SIBO) or history of intestinal polyps
2. Received any antibiotic in the last 30 days or known viral or bacterial illness in the last 30 days
3. Any NSAID use in the last 14 days
4. History of an autoimmune disease (including diabetes, autoimmune hepatitis, primary sclerosing cholangitis, thyroiditis, psoriasis or juvenile idiopathic arthritis)
5. Any condition that in the opinion of the PI will prevent the research participant from taking part in this study

Phase II - Longitudinal Study of Participants with CD

Inclusion Criteria:

1. Age criteria: > 1 year to < 22 years of age
2. Diagnosis of Crohn's disease with:

   1. Luminal inflammation (ulcerations in ileum and/or colon visible by ileocolonoscopy) and
   2. Endoscopic evidence of active Crohn's disease (up to 90 days prior to starting anti-TNF) OR if no colonoscopy within 90 days then fecal calprotectin ≥250 µg/g or fecal lactoferrin >10 µg/g (<90 days from starting anti-TNF)
3. Anti-TNF naïve
4. Starting infliximab or adalimumab (or either biosimilar)
5. Permission of parent/guardian and assent or consent of research participant

Exclusion Criteria:

1. Crohn's disease limited to esophagus, stomach, duodenum or jejunum
2. Prior treatment with infliximab, adalimumab, certolizumab or golimumab
3. Known diagnosis of Ulcerative colitis (UC) or inflammatory bowel disease-unspecified (IBD-U)
4. Active or prior evidence of internal (abdominal/pelvic) penetrating fistula(e)
5. Active intra-abdominal abscess or perianal abscess
6. Active Clostridium difficile infection or other known enteric infection in last 2 weeks
7. Current ileostomy or colostomy, extensive small bowel resection, ileoanal pouch or short bowel syndrome
8. History of autoimmune disease (including autoimmune hepatitis, primary sclerosing cholangitis, thyroiditis, psoriasis or juvenile idiopathic arthritis)
9. Contraindications to MRI scanning, such as metal implants/non-compatible medical devices or medical conditions
10. Any condition that in the opinion of the PI will prevent the research participant from taking part in this study

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Potential IBD participants will be recruited through the Division of Gastroenterology at each participating site.
  Healthy volunteers will be recruited from through direct advertising methods approved by the IRB and formal local databases intended for recruitment.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Sustained Deep Remission | 1 year
  Sustained Deep Remission, defined as meeting all of the following at 1 year (check all that apply):
  * no wPCDAI score of ≥12.5 on two consecutive visits between week 30-52
  * wPCDAI at week 52 is <12.5
  * off prednisone between weeks 30-52
  * endoscopic remission (SES-CD<3)

SECONDARY OUTCOMES:
End of Induction Outcomes: Clinical Response | Week 16
  Improvement of >17.5 points from baseline wPCDAI and/or Week 16 wPCDAI= <12.5 points
End of Induction Outcomes: Clinical Remission | Week 16
  wPCDAI <12.5 at Week 16
End of Induction Outcomes: Steroid Free Clinical Remission | Week 16
  wPCDAI <12.5 and off prednisone by Week 16
End of Induction Outcomes: Fecal Biochemical Response | Week 16
  Fecal calprotectin improved >50% from baseline stool (+/- 30 days from Week 16)
End of Induction Outcomes: Fecal Biochemical Remission | Week 16
  Fecal calprotectin <250µg/g at Week 16 (+/- 30 days)
End of Induction Outcomes: Blood CRP Biochemical Remission | Week 16
  CRP <0.5 mg/dL at Week 16
End of Induction Outcomes: Blood CD64 Biochemical Remission | Week 16
  nCD64 <4.5 at Week 16
Week 52 Outcomes: Endoscopic Response | 1 year
  50% reduction in SES-CD score from baseline SES-CD (if performed)
Week 52 Outcomes: Endoscopic Remission | 1 year
  SES-CD <3
Week 52 Outcomes: Minimal Endoscopic Activity | 1 year
  SES-CD <6 with no individual SES-CD subscore >1
Week 52 Outcomes: Complete Intestinal Healing | 1 year
  SES-CD = 0
Week 52 Outcomes: Sustained, Steroid-free Clinical Remission | 1 year
  wPCDAI <12.5 for all visits from weeks 30-52, off prednisone
Week 52 Outcomes: Clinical Remission | 1 year
  wPCDAI <12.5 and off prednisone at last study visit
Week 52 Outcomes: Clinical Remission and Endoscopic Response | 1 year
  wPCDAI <12.5 at week 52 and SES-CD>50% reduction from baseline
Week 52 Outcomes: Clinical Remission and Minimal Endoscopic Activity | 1 year
  wPCDAI <12.5 at week 52 and SES-CD<6 with no individual SES-CD subscore >1
Week 52 Outcomes: Treatment Response | 1 year
  continues on anti-TNF without surgery, hospitalization and off prednisone by week 16
Week 52 Outcomes: Transmural ileal healing | 1 year
  ileum subscore stage 0 (score = 0) or stage 1 (score 1-3)
Week 52 Outcomes: Transmural colonic healing | 1 year
  all segments of colon subscore stage 0 (score=0) or stage 1 (score 1-3)
Week 52 Outcomes: Total Bowel Transmural healing | 1 year
  total ileum and colonic subscore is not greater than stage 1 on either individual score
Week 52 Outcomes: Fecal Biochemical Remission | 1 year
  fecal calprotectin <250 µg/g at week 52
Week 52 Outcomes: Deep Fecal Biochemical Remission | 1 year
  fecal calprotectin <150 µg/g at week 52
Week 52 Outcomes: CRP Biochemical Remission | 1 year
  CRP <0.5 mg/dL at week 52
Week 52 Outcomes: CD64 Biochemical Remission | 1 year
  nCD64 <4.5 at week 52
Week 52 Outcomes: PGA Remission | 1 year
  physician-rated PGA is quiescent and subject is off prednisone

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Minar, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Velez Lopez A, Waddell A, Antonacci S, Castillo D, Santucci N, Ollberding NJ, Eshleman EM, Denson LA, Alenghat T. Microbiota-derived butyrate dampens linaclotide stimulation of the guanylate cyclase C pathway in patient-derived colonoids. Neurogastroenterol Motil. 2023 Dec;35(12):e14681. doi: 10.1111/nmo.14681. Epub 2023 Sep 22. PMID 37736865